CLINICAL TRIAL: NCT01405144
Title: Phase III Comparative Study About the Use of 5% 5-fluorouracil Cream Versus Its Utilization as Agent for Sequential Superficial Peeling in the Treatment of Advanced Photoaging
Brief Title: 5fluorouracil for Advanced Photoaging
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Edileia Bagatin, Universidade Federal de Sao Paulo - Dermatology Department
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Carol2011
Record Dates: First submitted 2011-07-05; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-05

CONDITIONS: Photoaging; Actinic Keratosis
Keywords: Photoaging; Actinic keratosis; 5-fluoruracil; Carcinogenesis
MeSH Terms: conditions — Keratosis, Actinic; Carcinogenesis | interventions — Therapeutics; Cosmetics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5% 5-fluoruracil cream (Active Comparator): 30 patients will use 5% 5-fluoruracil cream, twice a day, during 3 weeks, in one randomized forearm
  Interventions: Drug: 5-fluoruracil
- 5% 5-fluoruracil peeling (Active Comparator): The same 30 patients will be submitted to 4 applications of 5% 5-fluoruracil superficial peeling in the other forearm
  Interventions: Procedure: 5-fluoruracil

INTERVENTIONS:
Drug: 5-fluoruracil — 5% 5-fluoruracil cream, twice a day, during 3 weeks
  Other Names: Topical treatment
  Arms: 5% 5-fluoruracil cream
Procedure: 5-fluoruracil — The same 30 patients will be submitted to 4 weekly application of superficial peeling using 5% 5-fluoruracil in propyleneglycol as vehicle. The applications will be performed by physician (one of the co-investigators)
  Other Names: Cosmetic procedure
  Arms: 5% 5-fluoruracil peeling

SUMMARY:
It is well known the efficacy of 5% 5-fluoruracil for multiple and superficial actinic keratosis (AKs)treatment. Recently its additional benefit for advanced and severe photoaging while treating Aks was reported.

The aim of this study is to compare the efficacy and safety of the two modalities of 5% 5-FU use for forearms photoaging.

DETAILED DESCRIPTION:
The use of 5% 5-fluorouracil (5-FU) cream, twice a day, during 3 weeks represents a classic treatment for multiple and superficial AKs. The main adverse event is the severe skin irritation leading to interruption of the treatment in some cases. In the last decade a superficial pulse-peeling using it as agent in sequential applications was described. This modality of treatment has been demonstrated efficacy and better tolerability.

The improvement of the overall aspect of photodamaged skin is observed while treating multiple AKs.

There are no comparative study between the two types of 5% 5-FU use. So that is the purpose of our clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Men and women, aged from 50 to 75 anos;
2. Phototype I a III (Fitzpatrick Classification);
3. Advanced photoaging on forearms, with multiple superficial actinic keratosis;
4. Agreement with no sun exposure during the study and
5. Agreement with study conditions,capacity to understand and follow the orientations and form consent signature.

Exclusion Criteria:

1. Topical treatment with:

   * tretinoin in the last 6 months ;
   * other retinoids, alpha-hydroxyacids, poli-hydroxyacids, beta-hydroxyacids and ascorbic acid in the last 3 months;
2. Treatment by chemical peeling, microdermabrasion and non-ablative laser in the last 3 months;
3. Treatment with systemic retinoid in the last 6 months ;
4. Chemotherapy in the last 3 months;
5. Hypersensibility to parabens;
6. Infectious or inflammatory dermatosis on forearms;
7. Clinical evidence of immunosuppression and
8. Presence of photodermatosis

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-09 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Change in Photographic Evaluation | 0, 60, 180 days
  Photographic blinded evaluation by two independent observers, comparing modifications of forearms skin overall aspect before and after 60 and 180 days of the treatments. The following 5 point scale will be used: -2=much worse; -1=worse; 0=inlatered; 1=better, 2= much better
Change in Microscopic Evaluation | 0, 180 days
  Skin biopsies will be performed and coloration by hematoxilin-eosin, Verhoeff, Tricromio Masson , Picrosirius and biomarkers (p53, bcl2, collagen 1)will be used. The modifications on corneal layer and epidermal thickness, dermal elastotic material and collagen deposition and biomarkers expression will be evaluated by digital quantitative analysis, comparing the findings before (day 0) and after (day 180)treatments.

SECONDARY OUTCOMES:
Inflammatory Skin Reaction | 30 day
  Comparison between treatments on inflammatory skin reaction will be performed by expression of interleucin-1, using immunohistochemistry
Occurence and Evaluation of Adverse Events | 30, 60, 180 days
  Predictable and unpredictable side effects and their intensity related by patient and/or observed by investigator will be analized and compared between the treatments
Change in Patient Opinion | 0, 30, 60, 180 days
  Patient opinion concerning modification on forearms skin overall aspect, using a 5 point scale: -2=much worse; -1=worse; 0=inaltered; 1=better, 2= much better, comparing day 0 to 60, 60 to 180 and 0 to 180.
Change in Investigator Clinical Evaluation | 0, 30, 60, 180 days
  Investigator efficacy evaluation through actinic keratosis counting, on days 0, 30, 60 and 180 as weel as modification on forearms skin overall aspect. That will be performed by comparision of skin examination on days 60 and 180 to photography captured on days 0 and 60, i.e, 0 to 60, 60 to 180 and 0 to 180, using a 5 point scale: -2=much worse; -1=worse; 0=inaltered; 1=better, 2= much better
Change in Forearm Photoaging Classification | 0, 60, 180 days
  A classification will be created and validated by investigators and five independent observers previously to classify forearm photoaging. After validation it will be applied to study subjects on days 0, 60 and 180 to evaluate modification on the forearm photoaging grade for each tretament.

CONTACTS AND LOCATIONS:
Overall Officials: Ediléia Bagatin, PhD, Study Chair — Professor
Locations (1):
- Edileia Bagatin, São Paulo, São Paulo, Brazil